CLINICAL TRIAL: NCT04438720
Title: Bioequivalence of Extended Release Nifedipine Tablets in Healthy Chinese Subjects: A Single-dose and Two-period Crossover Study
Brief Title: Bioequivalence of Extended Release Nifedipine Tablets in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cao Yu (Other)
Responsible Party: Sponsor-Investigator, Cao Yu, Director, Head of Phase I clinical research center, Principal Investigator, Clinical Professor., The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Awk-2019-BE-03
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Therapeutic Equivalency
Keywords: Extended Release Nifedipine Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Release Nifedipine Tablets（Adalat® GITS） (Active Comparator): Extended Release Nifedipine reference formulation at a single dose of 30 mg
  Interventions: Drug: Extended Release Nifedipine Tablets 30 mg (Adalat® GITS)
- Extended Release Nifedipine Tablets (Experimental): Extended Release Nifedipine test formulation at a single dose of 30 mg
  Interventions: Drug: Extended Release Nifedipine Tablets 30 mg

INTERVENTIONS:
Drug: Extended Release Nifedipine Tablets 30 mg — The subjects randomly received single oral administration of extended release nifedipine tablets 30 mg.
  Arms: Extended Release Nifedipine Tablets
Drug: Extended Release Nifedipine Tablets 30 mg (Adalat® GITS) — The subjects randomly received single oral administration of extended release nifedipine tablets 30 mg.
  Arms: Extended Release Nifedipine Tablets（Adalat® GITS）

SUMMARY:
According to the relevant provisions of bioequivalence test, nifedipine sustained-release tablets (test preparation, t, 30mg / tablet) provided by Guangzhou bostao controlled release pharmaceutical Co., Ltd. were compared with Adalat ® GITS (reference preparation, R, 30mg / tablet) produced by Bayer Pharma AG to evaluate the bioequivalence of single dose in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged 18-45.
* The body mass index is in the range of 18.6-28.5 kg/m2 (including the critical value). The weight of male is not less than 50.0 kg, and that of female is not less than 45.0 kg.
* The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: Vital signs, physical examination, blood routine, blood biochemistry, urinalysis, pregnancy test for female, serological tests for hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), and syphilis virus, 12 lead ECG, breath test for alcohol, drug abuse test.
* The subjects have no family planning within 3 months and could select contraceptive method.
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.

Exclusion Criteria:

* Being allergy to the study medications, smoking, alcohol abuse.
* Participation in another clinical trial within 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-09-09 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 60 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 60 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 60 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 60 days
  Collection of adverse events
Incidence of abnormal blood pressure | 60 days
  Monitor both systolic and diastolic blood pressure
Incidence of abnormal temperature | 60 days
  Monitor the temperature
Incidence of abnormal pulse | 60 days
  Temperature the pulse
Incidence of abnormal electrocardiogram waveform | 60 days
  Electrocardiogram inspection

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China